CLINICAL TRIAL: NCT03144869
Title: Feasibility and Acceptability of Physical Activity Monitoring as an Educational Tool in the Management of Paediatric Type 1 Diabetes
Brief Title: Physical Activity Monitoring Paediatric Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Hallam University (Other)
Collaborators: Sheffield Children's NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Helen Quirk, Principal Investigator, Sheffield Hallam University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CA16015
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: type 1 diabetes mellitus; physical activity; children; constant glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical activity monitor only (Experimental): Children will wear a Runscribe accelerometer for two weeks. Runscribe is a small inertial sensor (weight 15g, size 35x25x7.5 mm). It can be attached to the body in several positions (wrist, waist, sacrum, chest, thigh, foot) and is used for monitoring movement. Runscribe does not beep, flash or have a visual display. It will not provide PA feedback to the individuals in real-time, only via a researcher after the data has been downloaded. In this study, we are not wishing to influence children's behaviour by providing PA feedback in real-time. We are trying to establish whether PA monitoring is feasible and acceptable - and further research could go on to explore the use of real-time PA feedback as an educational technique.
  Phase 1 findings will help to determine: i) method of monitor distribution to participants (post, clinic or in-person), ii) preferred wear position.
  Interventions: Behavioral: physical activity monitor and feedback
- physical activity monitor plus constant glucose monitor (Experimental): Children using a personal constant glucose monitor (CGM) or CGM on loan from clinic as part of clinical care will be approached for Arm 2. These children will wear Runscribe at the same time as a CGM. Runscribe and CGM worn over the same 2 week period.
  Interventions: Behavioral: physical activity monitor and feedback

INTERVENTIONS:
Behavioral: physical activity monitor and feedback — Children will wear a Runscribe accelerometer for two weeks (children in Arm 2 will also wear a CGM). Runscribe will measure activity levels. Activity data will be downloaded by a researcher, analysed and graphs of daily activity levels prepared. At the child's next routine clinic appointment, child and parent will have 1:1 session with researcher acting as 'physical activity champion'. Session content will be informed by Phase 1, but will involve educational support around PA (including barriers and facilitators to participation) and individualised feedback on PA level). Individualised feedback will involve review of daily PA graphs - addressing times of high and low activity levels. For participants in Arm 2, there will also be review of daily line graphs showing BG trends. As part of standard clinical care, CGM data gets downloaded at routine clinic appointments and is visible on the patient's clinic notes in daily graph form.

SUMMARY:
Physical activity (PA) can have positive health outcomes for children with type 1 diabetes (T1DM), yet being physically active can have unwanted side effects due to fluctuations in blood glucose (BG) level. Children and parents need support to help understand the relationship between PA and BG level, and how to use PA as a vehicle to better manage the condition. Using PA monitoring could help HCPs raise awareness about PA, discuss PA and facilitate diabetes management. This research will explore the feasibility and acceptability of PA monitoring as a clinical tool to help the management of paediatric T1DM.

DETAILED DESCRIPTION:
Physical activity (PA) can have positive health outcomes for children with type 1 diabetes (T1DM) such as improved diabetes control, lipid profile and body composition, yet activity levels are low. The unpredictable nature of children's everyday activity causes fluctuations in blood glucose (BG) level. Low and high BG level are side-effects of PA, have significant symptoms and can cause a range of chronic complications. Parents typically have responsibility for diabetes management in preadolescent children and perceive PA as a challenge due to constant concerns about BG levels (Quirk et al., 2015).

Children and parents need support to help understand the relationship between PA and BG control and how to use PA as a vehicle through which to better manage the condition. T1DM healthcare professionals (HCPs) perceive a lack of i) competence, ii) confidence and iii) time to provide PA advice and education in the clinical setting. HCPs perceive a need for evidence-based resources to facilitate PA discussion, education and promotion (Quirk et al., 2015). Physical activity monitoring is already a widely recognised and accepted tool, with potential utility in paediatric diabetes.

One such approach could be that HCPs graphically convey children's PA levels and use this to raise awareness and promote discussion about daily PA level. In those using constant glucose monitoring devices, daily BG values could be graphically documented to help explain the relationship between PA and BG level. These devices have shown acceptability among children with T1DM. However, whether they can facilitate PA discussion and education is unknown.

This research will explore parents, children and HCPs' perceptions of PA monitoring in clinical practice. A PA monitoring programme will be developed, implemented in a small cohort of children with T1DM and evaluated for feasibility and acceptability. In the future, 'physical activity clinical champions' could be trained to use activity monitoring for PA education and promotion in clinic settings.

ELIGIBILITY:
Inclusion Criteria:

* Arm 1 Children with type 1 diabetes Aged 7-11 years (age range may be increased to 6-12 years if recruitment is problematic) Diagnosed with type 1 diabetes for at least 12 months Consenting primary caregiver Willingness of child and parent for the child to wear activity monitor
* Arm 2 Children with type 1 diabetes using a personal CGM OR CGM on loan from clinic as part of clinical care Aged 7-11 years (age range may be increased to 6-12 years if recruitment is problematic) Diagnosed with type 1 diabetes for at least 12 months Consenting primary caregiver Willingness of child and parent for the child to wear an activity monitor

Exclusion Criteria:

-

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Recruitment | During recruitment (0 months)
  Recruitment will be recorded during the recruitment period as the number of eligible participants that consented to participate. The following data will be assessed: number meeting eligibility criteria, reasons for ineligibility, number consenting and reasons for non-participation; demographic profile of participating and nonparticipating (e.g., to assess inclusion of ethnic minority and hard-to-reach groups), and withdrawals (with reasons where available).
Adherence | At follow-up (~3 months)
  Adherence will refer to the proportion of participants who adhere to the activity monitoring protocol (meet the valid wear-time protocol) and proportion of participants who attend all scheduled activity monitoring sessions with the researcher. Adherence will be monitored by the researcher at baseline, follow-up and throughout the intervention.
Retention | At follow-up (~3 months)
  Retention rate will be defined as the number of participants completing the intervention, including all follow-up data collection (follow-up and interview) compared to the number started. Retention will be recorded by the researcher at follow-up and interview.
Data completion | At baseline (0 months) and follow-up (~3 months)
  Data completion rate is determined by recording the proportion of participants who complete the outcome measures at baseline and follow-up. To assess data completion, completion of questionnaire measures will be recorded at baseline and follow-up (complete and partial or non-completion with reasons, time to complete). The feasibility of gathering routinely collected data available in patients' clinic notes at baseline and follow-up will be assessed. Feasibility of collecting observational data in this way will be determined if >85% of our sample have complete clinical records available. Data completion will be recorded by the researcher at baseline and follow-up.
Occurrence of adverse events | At baseline (0 months), during intervention (0-3 months) and at follow-up (~3 months)
  ccurrence of adverse events related to the intervention (e.g., severe hypoglycaemia, accident or injury) will be assessed by reviewing patient notes and patient self-report.
Acceptability | At follow-up (~3 months)
  User acceptability of research and intervention processes will be assessed by interview with children and parents. Interviews will explore acceptability of i) recruitment, ii) outcome measures, iii) participant burden, iv) the activity monitor and v) feedback sessions to determine appropriateness of the intervention for use in a future trial and clinical practice. Interviews will explore perceptions of change. Interviews will be conducted by a member of the research team who is experienced in qualitative research and who, ideally, has had no direct involvement with the intervention implementation.

SECONDARY OUTCOMES:
Demographics | At baseline (0 months)
  A questionnaire developed specifically for this study that asks parents to report: child's age, child's ethnic background, use of glucometer/constant glucose monitor, method of insulin delivery, parental occupation, parental education, and total family income per year.
Clinical information | At baseline (0 months) and follow-up (~3 months)
  Clinical information will be collected from the participant's electronic clinic notes. These data collection methods are non-invasive (glycaemic control, insulin dosage, height and weight measurements - measured as routine at every clinic appointment- will be taken from the child's clinic notes, with permission). The researcher will ask clerical staff at the participating centre to complete a spreadsheet with the information for each consenting participant at baseline and follow-up. Data extracted will include: Height, Weight, Glycaemic control (HbA1c), Insulin dosage, Frequency of severe hypoglycaemia, Method of insulin delivery. This data is measured by trained nurses as standard at all routine clinic appointments. The researcher will ask for the data collected at the corresponding clinic appointment.
Parental self-efficacy for diabetes management | At baseline (0 months) and follow-up (~3 months)
  Parental self-efficacy for diabetes management will be assessed using the self-efficacy for diabetes scale (Streisand et al., 2005). It contains 22 parenting tasks associated with diabetes management, and parents rate their confidence with performing each task on a 5-point scale (1-Very sure I can't to 5-Very sure I can), indicating how much they believe they can or cannot do what is asked now. Higher scores indicate greater parental self-efficacy.
Parental fear of hypoglycaemia | At baseline (0 months) and follow-up (~3 months)
  Parental fear of hypoglycaemia will be assessed using the parents' Hypoglycemia Fear Survey (PHFS) (Gonder-Frederick et al., 2011). The PHFS is comprised of a 10-item behaviour (B) subscale and a 15-item worry (W) subscale. Higher scores indicate greater fear of hypoglycaemia. HFS-B items describe behaviours performed in order to avoid hypoglycaemic episodes and/or their negative consequences (e.g., by limiting exercise or physical activity). HFS-W items ask about specific concerns about hypoglycaemic episodes (e.g., episodes occurring during sleep, or having an accident). Higher scores indicate greater fear of hypoglycaemia. Research shows that the PHFS can provide reliable self-report of parental fear of hypoglycaemia (Gonder-Frederick et al., 2011). It also asks parents to report the number of severe hypoglycaemia episodes their child has experienced in the past 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Children's Hospital NHS Foundation Trust, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Streisand R, Swift E, Wickmark T, Chen R, Holmes CS. Pediatric parenting stress among parents of children with type 1 diabetes: the role of self-efficacy, responsibility, and fear. J Pediatr Psychol. 2005 Sep;30(6):513-21. doi: 10.1093/jpepsy/jsi076. Epub 2005 Mar 3. PMID 16055489
- [Background] Gonder-Frederick L, Nyer M, Shepard JA, Vajda K, Clarke W. Assessing fear of hypoglycemia in children with Type 1 diabetes and their parents. Diabetes Manag (Lond). 2011;1(6):627-639. doi: 10.2217/DMT.11.60. PMID 22180760